CLINICAL TRIAL: NCT01818505
Title: The Influence of Antiphospholipid Antibodies on the Relationship Between Hyperurecemia, Gout and Metabolic Syndrome
Acronym: URIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: URIC
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Antiphospholipid Syndrome; Endothelial Dysfunction; Hyperuricemia; Gout; Metabolic Syndrome
Keywords: antiphospholipid syndrome; gouty arthritis; Hyperuricemia; metabolic syndrome; osteoarthritis; cardiovascular co-morbidities
MeSH Terms: conditions — Antiphospholipid Syndrome; Hyperuricemia; Gout; Metabolic Syndrome; Arthritis, Gouty; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Gouty arthritis: Patient with gouty arthritis
- Asymptomatic hyperuricemia: Patient with asymptomatic hyperuricemia
- OA without hyperuricemia: Patient of osteoarthritis but without hyperuricemia and gout

SUMMARY:
Patients with hyperuricemia were confirmed to have higher risks of cardiovascular disease, but the exact mechanism remained to be elucidated. Many connective tissue diseases such as rheumatoid arthritis are often associated with antiphospholipid antibodies-associated endothelial impairment. In the present study, the investigators will analyze the presence of antiphospholipid antibodies in the serum of the patients with gout/asymptomatic hyperuricemia, with a comparison to the patients of osteoarthritis but without hyperuricemia and gout. The investigators expect to find a correlation between these pathogenic antibody and those cardiovascular co-morbidities.

DETAILED DESCRIPTION:
Patients with hyperuricemia were confirmed to have higher risks of cardiovascular disease, but the exact mechanism remained to be elucidated. Many connective tissue diseases such as rheumatoid arthritis are often associated with antiphospholipid antibodies-associated endothelial impairment. In the present study, we'll analyze the presence of antiphospholipid antibodies in the serum of the patients with gout/ asymptomatic hyperuricemia, with a comparison to the patients of osteoarthritis but without hyperuricemia and gout. We expect to find a correlation between these pathogenic antibody and those cardiovascular co-morbidities.

Patient eligibility：

1. Patients with gout
2. Patients with asymptomatic hyperuricemia
3. Patients of osteoarthritis but without hyperuricemia and gout Exclusion Criteria： Patients younger than 20 years old

ELIGIBILITY:
Inclusion Criteria:

1. Patient with gouty arthritis
2. Patient with asymptomatic hyperurecemia
3. Patient of osteoarthritis but without hyperuricemia and gout

Exclusion Criteria:

1.Patient younger than 20 y/o.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
development of metabolic syndrome or cardiovascular events | 36 months

SECONDARY OUTCOMES:
Acute myocardial infarct or stroke | 36 months or more

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Min Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Dou-Liou City, Yun-Lin County, Taiwan